CLINICAL TRIAL: NCT01833169
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 1 - BKM120 for Patients With PI3K-activated Tumors
Brief Title: BKM120 for Patients With PI3K-activated Tumors
Acronym: SIGNATURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120ZUS40
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: PI3K Pathway Activated Tumors
Keywords: Solid tumor; malignancy; hematologic malignancy; PI3K pathway activation; P13K activated tumors; BKM120; signature; AML; acute myelogenous leukemia; cervical; ovarian; hepatobiliary; buparlisib
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Leukemia, Myeloid, Acute | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 (Experimental): BKM120 100 mg (oral gelatine capsules) was administered orally once daily starting from cycle 1 day 1 and will be dosed continuously every day for each 28- day cycle
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — BKM120 100 mg (oral gelatine capsules) was administered orally once daily starting from cycle 1 day 1 and will be dosed continuously every day for each 28-day cycle

SUMMARY:
The purpose of this signal seeking study was is to determine whether treatment with BKM120 demonstrates sufficient efficacy in select pathway-activated solid tumors and/or hematologic malignancies to warrant further study.

ELIGIBILITY:
Inclusion Criteria:

* Patient had a confirmed diagnosis of a solid tumor or hematological malignancy with the exception of endometrial cancer, glioblastoma, nonsmall cell lung cancer, prostate cancer or breast cancer.
* Patient's tumor was evaluated and pre-identified to have activation of the PI3K pathway, at a CLIA certified laboratory
* Patient must have received at least one prior treatment for recurrent metastatic and /or locally advanced disease and for whom no standard therapy options was anticipated to result in a durable remission.
* Patient must have had progressive and measurable disease as per RECIST 1.1. or other appropriate hematological guidelines
* Patient had an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

Patient had received previous treatment with BKM120 Patient had symptomatic CNS metastases Patient had mood disorder as outlined in Section 5 Patient had received chemotherapy or other anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (59):
  - Arizona Oncology Associates HOPE Division, Phoenix, Arizona
  - Arizona Oncology Associates PC- HAL, Sedona, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Sarcoma Oncology Center, Santa Monica, California
  - Rocky Mountain Cancer Centers RMCC - Aurora, Greenwood Village, Colorado
  - Whittingham Cancer Center Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates The Norwich Cancer Center, Norwich, Connecticut
  - Florida Cancer Specialists Dept of Oncology (2), Fort Myers, Florida
  - Florida Hospital Cancer Institute FL Hosp. Cancer Instit., Orlando, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Illinois Cancer Care P.C. IL. Cancer Care, Peoria, Illinois
  - Illinois Cancer Care P.C., Peoria, Illinois
  - Cancer Treatment Centers of America Southwestern Regional Med. Ctr, Schaumburg, Illinois
  - Northern Indiana Cancer Research Consortium No. Indiana Cancer Res., South Bend, Indiana
  - University of Iowa Hospitals & Clinics Regulatory Contact 2, Iowa City, Iowa
  - Eastern Maine Medical Center Research Center SC, Bangor, Maine
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - Michigan Medicine University of Michigan Int. Medicine Oncology, Ann Arbor, Michigan
  - Cancer and Hematology Centers of West Michigan Dept. of Oncology, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, P.A. Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Nebraska Cancer Specialists Oncology Hematology West, Omaha, Nebraska
  - Comprehensive Cancer Centers, Las Vegas, Nevada
  - Hematology Oncology Associates of Northern New Jersey PA Regional Cancer Care Assoc., Morristown, New Jersey
  - Cancer Center at Presbyterian, Albuquerque, New Mexico
  - New York Oncology Hematology NY Onc Hem, Albany, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - University of N C at Chapel Hill Physician Office Building, Chapel Hill, North Carolina
  - Duke University Medical Center Seeley G. Mudd Bldg., Durham, North Carolina
  - Cleveland Clinic Foundation Cleveland Clinic (19), Cleveland, Ohio
  - Mid Ohio Oncology/Hematology Mark H. Zangmeister Center, Columbus, Ohio
  - Bend Memorial Clinic Bend Mem. Clinic, Bend, Oregon
  - Northwest Cancer Specialists Compass Oncology (36), Portland, Oregon
  - Oregon Health and Science University Oregon Health & Science U (56), Portland, Oregon
  - Salem Health, Salem, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - West Penn Allegheny Oncology Network, Natrona Heights, Pennsylvania
  - University of Pittsburgh Medical Center UPMC, Pittsburgh, Pennsylvania
  - Abington Hematology Oncology Associates, Inc Abington Hem Onc Assoc (5), Willow Grove, Pennsylvania
  - Sanford University of South Dakota Medical Center Sanford Health, Sioux Falls, South Dakota
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - West Cancer Clinic, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology P A Round Rock, Dallas, Texas
  - Texas Oncology Sammons Cancer Center Sammons Cancer Center (10), Dallas, Texas
  - Texas Oncology, P.A. Texas Oncololgy, P.A. (8), Fort Worth, Texas
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Cancer Care Centers of South Texas HOAST CCC of So. TX-San Antonio (3), San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Virginia Cancer Specialists Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Research Center at Roanoke Neurological Center McKesson Specialty Care, Roanoke, Virginia
  - Kadlec Clinic Hematology and Oncology Kadlec Clinic Hematology & Onc, Kennewick, Washington
  - Northwest Medical Specialties Hematology/Oncology, Tacoma, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to informed consent, patient was pre-identified to have activation of the P13K pathway confirmed via Genomic Profiling Report and whose disease had progressed on or after standard treatment
Period: Overall Study
Arm/Group | BKM120
Started | 146
Consented to be Followed for Survival | 128
Completed | 0
Not Completed | 146
Not completed — Disease Progression | 99
Not completed — Adverse Event | 33
Not completed — Withdrawal by Subject | 9
Not completed — Death | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | BKM120
Number analyzed (Participants) | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 61
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 130
  Black | 7
  Asian | 3
  Other | 6
ECOG Grade [Number; unit: participants] — ECOG Scoring: 0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work, 2=Ambulatory and capable of all self-care but unable to carry out any work activities.
  Up and about more than 50% of waking hours, 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, Cannot carry on any self-care. Totally confined to bed or chair, 5= Dead
  participants
    Grade 0 | 54
    Grade 1 | 91
    Grade 2 | 1
Protocol pre-defined gene mutation (by local labs) [Number; unit: participants]
  PIK3CA gene mutation | 74
  PTEN gene mutation | 60
  PIK3CA amplification | 19
  PIK3R1 gene mutation | 7
Prior Lines of Antineoplastic Medications [Median (Full Range); unit: Number of prior lines of treatment] | 3 [1 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Participant Clinical Benefit Response Rate
Description: Clinical benefit rate for patients with solid tumors will be assessed using RECIST 1.1 and will include responses of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) at >=16 weeks. For hematologic tumors other appropriate hematological response criteria was applied. Response criteria: CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm., PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study, PD= At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline
Time Frame: Week 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKM120
Number analyzed (Participants) | 146
percentage of participants | 15.1 [9.7 to 21.9]

2. Secondary Outcome: Overall Response of Partial Response (PR) or Greater. PR=at Least a 30% Decrease in the Sum of Diameters of Target Lesions, Taking as Reference the Baseline Sum Diameters
Description: Overall Response (OR) of Partial Response (PR) or greater is based on local investigator assessment. For patients with solid tumors, the assessment criteria will be RECIST 1.1 and will include responses of CR and/or PR. For hematologic tumors other appropriate hematological response criteria apply
Time Frame: baseline and every 8 weeks until disease progression or end of treatment, assessed up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BKM120
Number analyzed (Participants) | 146
percentage of patients | 1.4 [0.2 to 4.9]

3. Secondary Outcome: Progression-Free Survival - Number of Participants With an Event
Description: Progression free survival (PFS) is defined as the time from the date of first dose to the date of first documented disease progression or relapse or death due to any cause
Time Frame: Every 8 Weeks until death, assessed up to 24 months
Measure: Number; unit: participants
Arm/Group | BKM120
Number analyzed (Participants) | 146
participants
  participants with an event | 112
  participants censored | 34

4. Secondary Outcome: Progression-Free Survival (PFS)- Kaplan-Meier Estimates of PFS Timing in Months
Description: as for outcome 3
Time Frame: baseline up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 146
months | 1.9 [1.8 to 2.34]

5. Secondary Outcome: Progression-Free Survival (PFS)- Kaplan-Meier Estimates of PFS Rate in Percentages
Description: as for outcome 3
Time Frame: baseline up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKM120
Number analyzed (Participants) | 146
percentage of participants
  1 month | 88.4 [81.5 to 92.9]
  2 months | 43.8 [34.9 to 52.3]
  3 months | 39.4 [30.7 to 47.9]
  4 months | 20.4 [13.5 to 28.3]
  5 months | 20.4 [13.5 to 28.3]
  6 months | 14.1 [8.2 to 21.5]
  9 months | 5.8 [2.1 to 12.1]
  12 months | 2.9 [0.6 to 8.6]
  18 months | 1.4 [0.1 to 6.7]
  24 months | 0.0 [NA to NA] — confidence interval could not be determined because 0 patients had an event

6. Secondary Outcome: Overall Survival - Number of Participants With an Event
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause. If a patient is not known to have died, survival time will be censored at the date of the last contact
Time Frame: Every 8 Weeks until death, assessed up to 24 months
Measure: Number; unit: participants
Arm/Group | BKM120
Number analyzed (Participants) | 146
participants
  participants with an event | 110
  participants censored | 36

7. Secondary Outcome: Overall Survival (OS)- Kaplan-Meier Estimates of OS Timing in Months
Description: as for outcome 6
Time Frame: baseline up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 146
months | 6.3 [5.2 to 8.8]

8. Secondary Outcome: Overall Survival (OS)- Kaplan-Meier Estimates of OS Rate in Percentages
Description: as for outcome 6
Time Frame: baseline up to 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKM120
Number analyzed (Participants) | 146
percentage of participants
  1 month | 97.3 [92.8 to 99.0]
  2 months | 83.4 [76.2 to 88.5]
  3 months | 73.5 [65.5 to 80.0]
  4 months | 61.5 [53.0 to 68.9]
  5 months | 60.1 [51.6 to 67.6]
  6 months | 51.5 [43.0 to 59.4]
  9 months | 41.3 [33.2 to 49.3]
  12 months | 30.2 [22.6 to 38.1]
  18 months | 18.6 [11.9 to 26.4]
  24 months | 12.2 [5.0 to 22.7]
  30 months | 12.2 [5.0 to 22.7]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Treatment Last Visit (LPLV). All AEs reported I this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 30 months.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events field "number of deaths resulting from adverse events" all those deaths resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- BKM120: BKM120
Arm/Group | BKM120
Serious Adverse Events (participants affected / at risk) | 59/146
Other Adverse Events (participants affected / at risk) | 141/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=146)
Anaemia (Blood and lymphatic system disorders) | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Oesophageal perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 3
Bacteraemia (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 2
Pelvic abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Urinary tract infection bacterial (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Ammonia increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Psychotic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=146)
Anaemia (Blood and lymphatic system disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 51
Dry mouth (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 66
Vomiting (Gastrointestinal disorders) | 40
Fatigue (General disorders) | 72
Mucosal inflammation (General disorders) | 11
Oedema peripheral (General disorders) | 14
Urinary tract infection (Infections and infestations) | 12
Alanine aminotransferase increased (Investigations) | 27
Aspartate aminotransferase increased (Investigations) | 35
Blood alkaline phosphatase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 9
Lipase increased (Investigations) | 9
Weight decreased (Investigations) | 35
Decreased appetite (Metabolism and nutrition disorders) | 58
Dehydration (Metabolism and nutrition disorders) | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 40
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 12
Hyponatraemia (Metabolism and nutrition disorders) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 15
Headache (Nervous system disorders) | 13
Tremor (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 41
Confusional state (Psychiatric disorders) | 12
Depression (Psychiatric disorders) | 41
Insomnia (Psychiatric disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 24
Hypertension (Vascular disorders) | 9

LIMITATIONS AND CAVEATS:
Secondary objective: Duration of response was not analyzed due to low response rate observed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.